CLINICAL TRIAL: NCT00903175
Title: An Open-label, Multicenter Phase II Study to Compare the Efficacy and Safety of RAD001 as First-line Followed by Second-line Sunitinib Versus Sunitinib as First-line Followed by Second-line RAD001 in the Treatment of Patients With Metastatic Renal Cell Carcinoma.
Brief Title: Efficacy and Safety Comparison of RAD001 Versus Sunitinib in the First-line and Second-line Treatment of Patients With Metastatic Renal Cell Carcinoma
Acronym: RECORD-3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001L2202; 2009-011056-21 (EudraCT Number)
Record Dates: First submitted 2009-04-24; First posted 2009-05-18 (Estimated); Results first posted 2016-06-28 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-10

CONDITIONS: Renal Cell Carcinoma
Keywords: RAD001; everolimus; sunitinib; renal cell carcinoma; kidney cancer; metastatic renal cell cancer; advanced kidney cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Everolimus; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- everolimus 1L/sunitinib 2L (Experimental): everolimus First Line: 10 mg orally, once daily, (two 5 mg tablets), continuous treatment. sunitinib Second Line: 50 mg orally, once daily, 4 weeks on treatment followed by 2 weeks off (4/2)
  Interventions: Drug: everolimus; Drug: sunitinib
- sunitinib 1L/everolimus 2L (Active Comparator): sunitinib First Line: 50 mg orally, once daily, 4 weeks on treatment followed by 2 weeks off (4/2) everolimus Second Line: 10 mg orally, once daily (two 5 mg tablets), continuous treatment
  Interventions: Drug: everolimus; Drug: sunitinib

INTERVENTIONS:
Drug: everolimus — Everolimus was administered orally at 10 mg/day. Everolimus is formulated as tablets of 5 mg strength, blister-packed under aluminum foil in units of 10 tablets.
  Other Names: RAD001
Drug: sunitinib — Sunitinib was administered orally 50 mg daily, on a schedule of 4 weeks on/2 weeks off. Sunitinib was supplied as hard gelatin capsules of 12.5 mg, 25 mg, or 50 mg strength according to local practice.

SUMMARY:
This study assessed the efficacy and safety of first-line RAD001 followed by second-line sunitinib versus the opposite sequence: first-line sunitinib followed by second-line RAD001 for the treatment of patients with MRCC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced renal cell carcinoma.
2. Patients with at least one measurable lesion.
3. Patients with a Karnofsky Performance Status ≥70%.
4. Adequate bone marrow function.
5. Adequate liver function.
6. Adequate renal function.
7. Left ventricular ejection fraction (LVEF) ≥ lower limit of institutional normal (LLN)
8. Women of childbearing potential must have had a negative serum pregnancy test within 14 days prior to the administration of the study medication. Adequate contraception must be used while on study.

Exclusion Criteria:

1. Less than 4 weeks post-major surgery
2. Patients who had radiation therapy within 4 weeks prior to start of study treatment (palliative radiotherapy to bone lesions allowed within 2 weeks prior to study treatment start).
3. Patients in need for major surgical procedure during the course of the study
4. Patients with a serious non-healing wound, ulcer, or bone fracture
5. Patients with a history of seizure(s) not controlled with standard medical therapy
6. Patients who have received prior systemic treatment for their metastatic RCC
7. Patients who have previously received systemic mTOR inhibitors (sirolimus, temsirolimus, everolimus) or VEGF inhibitors. Note: History of adjuvant immunotherapy, vaccines or adjuvant sorafenib following localized surgical nephrectomy is acceptable.
8. Patients with a known hypersensitivity to RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus) or to its excipients Patients with a known hypersensitivity to RAD001 (everolimus) or other rapamycins or to its excipients
9. Patients with a known hypersensitivity to sunitinib or its excipients
10. History or clinical evidence of central nervous system (CNS) metastases. Note: Subjects who have previously-treated CNS metastases (surgery plus or minus radiotherapy, radiosurgery, or gamma knife) and meet all 3 of the following criteria are eligible:

    * Are asymptomatic and,
    * have had no evidence of active CNS metastases for ≥ 6 months prior to enrollment and,
    * have no requirement for steroids or enzyme-inducing anticonvulsants (EIAC)
11. Clinically significant gastrointestinal abnormalities including, but not limited to:

    * Malabsorption syndrome
    * Major resection of the stomach or small bowel that could affect the absorption of study drug
    * Active peptic ulcer disease
    * Inflammatory bowel disease
    * Ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation
    * History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment.
12. Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥160mmHg or diastolic blood pressure (DBP) of ≥ 95mmHg]
13. Patients receiving chronic systemic treatment with corticosteroids or another immunosuppressive agent
14. Patients with a known history of HIV seropositivity.
15. Patients with active bleeding.
16. Patients who have any severe and/or uncontrolled medical conditions or other conditions within the past 12 months that could affect their participation in the study such as:

    * Cardiac angioplasty or stenting, unstable angina pectoris, symptomatic peripheral vascular disease, symptomatic congestive heart failure (NYHA II, III, IV), myocardial infarction ≤ 6 months prior to first study treatment, serious uncontrolled cardiac arrhythmia, cerebrovascular accidents ≤ 6 months before study treatment start.
    * Prolongation of corrected QT interval (QTc) > 500 milliseconds (msecs).
    * Severally impaired lung function as defined as spirometry and DLCO that is 50% of the normal predicted value and/or 0^2 saturation that is 88% or less at rest on room air.
    * Poorly controlled diabetes as defined by fasting serum glucose >2.0 x ULN.
    * Any active (acute or chronic) or uncontrolled infection/disorders that impair the ability to evaluate the patient or for the patient to complete the study.
    * Liver disease such as chronic active hepatitis or chronic persistent hepatitis.
17. History of cerebrovascular accident (CVA) including transient ischemic attack (TIA).
18. History of pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months. Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible.
19. Patients who have a history of another primary malignancy and off treatment for ≤ 3 years
20. Female patients of child-bearing potential who are not using adequate birth control methods, or who are pregnant or breast feeding.
21. Patients who are using other investigational agents or who had received investigational drugs ≤ 2 weeks prior to study treatment start.
22. Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2009-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (81):
- United States (35):
  - University of Alabama at Birmingham/ Kirklin Clinic Comprehensive CancerCenter (1), Birmingham, Alabama
  - University of South Alabama / Mitchell Cancer Institute Dept. of Mitchell Cancer Inst., Mobile, Alabama
  - Highlands Oncology Group HighlandsOncGrp-Bentonville(2), Fayetteville, Arkansas
  - University of California San Diego - Moores Cancer Center Dept of Moores Cancer Ctr (5), La Jolla, California
  - University of California at Los Angeles Dept. of UCLA (3), Los Angeles, California
  - University of Colorado Dept. of Anschutz Cancer (2), Aurora, Colorado
  - Norwalk Hospital Norwlak SC, Norwalk, Connecticut
  - Georgetown University/Lombardi Cancer Center Dept.of Lombardi Cancer Ctr (2, Washington D.C., District of Columbia
  - Lynn Cancer Institute, Boca Raton, Florida
  - University of Miami SC, Miami, Florida
  - MD Anderson Cancer Center - Orlando Dept.ofMDACC-Orlando, Orlando, Florida
  - University Cancer & Blood Center, LLC Dept of NE GCC (2), Athens, Georgia
  - Georgia Health Sciences University Dept. of MCG, Augusta, Georgia
  - Summit Cancer Care, Savannah, Georgia
  - NorthwesternUniv.Med.School/Robert H. Lurie Comp.Cancer Ctr Dept.ofNorthwesternMemHospital, Chicago, Illinois
  - Loyola University Medical Center /Cardinal Bernardin Cancer Cardinal Bernardin Cancer (3), Maywood, Illinois
  - Crescent City Research Consortium, LLC SC, Metairie, Louisiana
  - VA Maryland Health Care Dept.of GreenbaumCancerCent(7), Baltimore, Maryland
  - Weinberg Cancer Institute at Franklin Square Hospital, Baltimore, Maryland
  - Billings Clinic Dept of Billings Clinic(2), Billings, Montana
  - Hackensack University Medical Center DeptofHackensackUniv.MedCtr., Hackensack, New Jersey
  - Cooper Cancer Center, Voorhees Township, New Jersey
  - Clinical Research Alliance, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center Dept. of MSKCC, New York, New York
  - SUNY - Upstate Medical University Div. of Hematology-Oncology, Syracuse, New York
  - University of North Carolina Dept. of LinbergerCancerCtr(3), Chapel Hill, North Carolina
  - Levine Cancer Institute Oncology, Charlotte, North Carolina
  - Duke University Medical Center Duke, Durham, North Carolina
  - University of Oklahoma Health Sciences Center Dept of OHSC, Oklahoma City, Oklahoma
  - St. Luke's Hospital and Health Network St Luke's Hospital (2), Bethlehem, Pennsylvania
  - The West Clinic Dept. of the West Clinic, Memphis, Tennessee
  - The Center for Cancer and Blood Disorders Dept. of The Ctr for C & BD(2), Fort Worth, Texas
  - East Texas Medical Center Cancer Institute, Tyler, Texas
  - Utah Cancer Specialists Dept.of Utah Cancer Spec. (3), Salt Lake City, Utah
  - Aurora Advanced Healthcare SC, Milwaukee, Wisconsin
- Argentina (4):
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
- Novartis Investigative Site, Woodville, South Australia, Australia
- Brazil (3):
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (8):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Saskatoon, Saskatchewan
- Novartis Investigative Site, Herlev, Denmark
- France (4):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Vandoeuvre-Les-Nancy Cede
- Germany (3):
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Weiden
- Hong Kong (2):
  - Novartis Investigative Site, Hong Kong, Hong Kong
  - Novartis Investigative Site, Shatin, New Territories, Hong Kong
- Italy (3):
  - Novartis Investigative Site, Arezzo, AR
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Chihuahua City, Chihuahua, Mexico
- Netherlands (2):
  - Novartis Investigative Site, Maastricht
  - Novartis Investigative Site, The Hague
- Novartis Investigative Site, Jesus Maria, Lima region, Peru
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Daejeon
- Spain (4):
  - Novartis Investigative Site, Elche, Alicante
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Lleida, Catalonia
- Taiwan (2):
  - Novartis Investigative Site, Niaosong Township, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan, ROC
- Novartis Investigative Site, Bangkok, Thailand
- Novartis Investigative Site, Istanbul, Turkey (Türkiye)
- United Kingdom (3):
  - Novartis Investigative Site, Bristol, Avon
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Nottingham

REFERENCES:
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Voss MH, Chen D, Reising A, Marker M, Shi J, Xu J, Ostrovnaya I, Seshan VE, Redzematovic A, Chen YB, Patel P, Han X, Hsieh JJ, Hakimi AA, Motzer RJ. PTEN Expression, Not Mutation Status in TSC1, TSC2, or mTOR, Correlates with the Outcome on Everolimus in Patients with Renal Cell Carcinoma Treated on the Randomized RECORD-3 Trial. Clin Cancer Res. 2019 Jan 15;25(2):506-514. doi: 10.1158/1078-0432.CCR-18-1833. Epub 2018 Oct 16. PMID 30327302
- [Derived] Knox JJ, Barrios CH, Kim TM, Cosgriff T, Srimuninnimit V, Pittman K, Sabbatini R, Rha SY, Flaig TW, Page RD, Beck JT, Cheung F, Yadav S, Patel P, Geoffrois L, Niolat J, Berkowitz N, Marker M, Chen D, Motzer RJ. Final overall survival analysis for the phase II RECORD-3 study of first-line everolimus followed by sunitinib versus first-line sunitinib followed by everolimus in metastatic RCC. Ann Oncol. 2017 Jun 1;28(6):1339-1345. doi: 10.1093/annonc/mdx075. PMID 28327953
- [Derived] Motzer RJ, Barrios CH, Kim TM, Falcon S, Cosgriff T, Harker WG, Srimuninnimit V, Pittman K, Sabbatini R, Rha SY, Flaig TW, Page R, Bavbek S, Beck JT, Patel P, Cheung FY, Yadav S, Schiff EM, Wang X, Niolat J, Sellami D, Anak O, Knox JJ. Phase II randomized trial comparing sequential first-line everolimus and second-line sunitinib versus first-line sunitinib and second-line everolimus in patients with metastatic renal cell carcinoma. J Clin Oncol. 2014 Sep 1;32(25):2765-72. doi: 10.1200/JCO.2013.54.6911. Epub 2014 Jul 21. PMID 25049330
- See also: Related Info — http://NovartisClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 238 patients were randomized to everolimus as 1st line followed by 2nd line sunitinib. All patients in this group were treated. 233 patients were randomized to the sunitinib as 1st line followed by 2nd line everolimus. However 2 of the 233 patients were not treated in this group.
Pre-assignment Details: The trial had a crossover design: first-line therapy until disease progression followed by second-line therapy until disease progression.Patients were randomized 1:1 to either everolimus-sunitinib or sunitinib-everolimus treatment sequence and were stratified by MSKCC risk criteria
Period: Period 1 - First Line
Arm/Group | Everolimus 1L/Sunitinib 2L | Sunitinib 1L/Everolimus 2L
Started | 238 | 231
Completed | 161 (Completed = Disease progression (completed 1L)) | 142 (Completed = Disease progression (completed 1L))
Not Completed | 77 | 89
Not completed — Adverse Event | 36 | 50
Not completed — Abnormal lab value(s) | 0 | 1
Not completed — Abnormal test procedure result(s) | 1 | 0
Not completed — Protocol Violation | 3 | 3
Not completed — Withdrawal by Subject | 8 | 12
Not completed — Administrative problems | 12 | 13
Not completed — Death | 17 | 10
Period: Period 2 - Second Line
Arm/Group | Everolimus 1L/Sunitinib 2L | Sunitinib 1L/Everolimus 2L
Started | 128 (139 from everolimus 1L planned to enter 2L period and cross over to sunitinib but only 128 did.) | 116 (130 from Sunitinib 1L planned to enter 2L period and cross over to everolimus but only 116 did.)
Completed | 79 (Completed = Disease progression - (completed 2L)) | 80 (Completed = Disease progression - (completed 2L))
Not Completed | 49 | 36
Not completed — Missing | 1 | 0
Not completed — Adverse Event | 16 | 20
Not completed — Withdrawal by Subject | 7 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Administrative problems | 19 | 9
Not completed — Death | 5 | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consists of all randomized patients. Following the intent-to-treat principle, patients are analyzed according to the treatment sequence and stratum they were assigned to at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus 1L/Sunitinib 2L | Sunitinib 1L/Everolimus 2L | Total
Number analyzed (Participants) | 238 | 233 | 471
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.36 (12.102) | 60.84 (11.627) | 61.10 (11.860)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 72 | 57 | 129
  Male | 166 | 176 | 342

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival First-Line (PFS 1-L)
Description: PFS_1L based on investigator assessment of radiology data by RECIST 1.0, was defined as the time from the date of randomization to the date of the first documented disease progression or death due to any cause during or after first-line treatment with everolimus or sunitinib. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: based on radiological assessments every 3 months until disease progression, start of another antineoplastic therapy or for any other reason up to 35 months
Population: The Full Analysis Set (FAS) consists of all randomized patients analyzed according to the treatment and stratum they were assigned to at randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus 1L/Sunitinib 2L | Sunitinib 1L/Everolimus 2L
Number analyzed (Participants) | 238 | 233
Months | 7.85 [5.55 to 8.25] | 10.71 [8.18 to 11.53]
Statistical Analysis 1: Comparison: Everolimus 1L/Sunitinib 2L vs Sunitinib 1L/Everolimus 2L; Test type: Non-Inferiority or Equivalence — Primary objective was to assess the non-inferiority of everolimus as compared to Sunitinib in terms of PFS-1L & was based on Bayesian methodology. If the estimated HR for PFS-1L had a value ≤ 1.1, non-inferiority of everolimus to Sunitinib would be declared. Non-inferiority of everolimus compared with Sunitinib as a first-line therapy was not achieved. The estimated HR for PFS-1L was 1.43 which did not satisfy the protocol-defined non-inferiority margin of a HR ≤ 1.1; Hazard Ratio (HR) = 1.43, 95% CI 2-sided [1.15 to 1.77]

2. Secondary Outcome: Progression-free Survival Combined (PFS-C)
Description: PFS-C (1L and 2L study drugs combined) was a composite endpoint which combined both lines of study treatment. It was defined as the time from the date of randomization to the first of the following: date of death due to any cause, or date of the first radiologically documented progression disease during or after the second-line treatment period for patients with a radiologically documented progression disease in the first-line treatment period and who had crossed-over to second-line treatment no more than 6 weeks after progression.
Time Frame: based on radiological assessments every 3 months until disease progression, start of another antineoplastic therapy or for any other reason up to about 56 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus 1L/Sunitinib 2L | Sunitinib 1L/Everolimus 2L
Number analyzed (Participants) | 238 | 233
Months | 21.68 [15.05 to 26.71] | 22.18 [16.03 to 29.83]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from date of randomization to date of death due to any cause. The analysis of OS included all deaths in the FAS regardless of when they were observed.
Time Frame: Every 2 months from randomization up to 3 years after last patient randomized
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus 1L/Sunitinib 2L | Sunitinib 1L/Everolimus 2L
Number analyzed (Participants) | 238 | 233
Months | 22.41 [18.60 to 33.28] | 29.47 [22.83 to 33.05]

4. Secondary Outcome: Overall Response Rate (ORR) - First -Line (1-L)
Description: ORR was defined as the number of participants with best overall response (BOR) of complete response (CR) or partial response (PR) and was based on investigator assessment of radiology data per RECIST. Participants with best overall response of 'Unknown' were treated as non-responders in the calculation of the ORR. Confirmed CR = at least two determinations of CR at least 4 weeks apart before progression. Confirmed PR = at least two determinations of PR or better at least 4 weeks apart before progression. CR required a disappearance of all target and non-target lesions. PR required at least a 30% decrease in the sum of the longest diameters of all target lesions, taking as a reference the baseline sum of the longest diameters. Radiological assessments : every 12 weeks until disease progression, the start of another antineoplastic therapy or for any other reason.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Everolimus 1L/Sunitinib 2L | Sunitinib 1L/Everolimus 2L
Number analyzed (Participants) | 238 | 233
percentage of participants
  Complete Response (CR) | 1 | 3
  Partial Response (PR) | 18 | 59
  Overall Response Rate (CR + PR) | 19 | 62

5. Secondary Outcome: Duration of Response (DoR) - First-Line (1-L)
Description: Duration of overall response (CR or PR) applies only to patients whose Best Overall Response (BOR) was Complete Response (CR) or Partial Response (PR) during the first-line treatment period. The start date was the date of first documented response (CR or PR) during the first-line treatment and the end date was the date of the event defined as the first documented progression or death due to underlying cancer during or after the same treatment line.
Time Frame: as for outcome 1
Population: The analysis population corresponds to the patients included in the Full analysis set (i.e. randomized patients analyzed according to the treatment and stratum they were assigned to at randomization) and who achieved a best overall response of CR or PR during the first-line treatment period.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus 1L/Sunitinib 2L | Sunitinib 1L/Everolimus 2L
Number analyzed (Participants) | 19 | 62
Months | 13.37 [8.3 to NA] — N/A = Data not estimable due to few number of patient at this time point | 17.25 [11.4 to NA] — N/A = Data not estimable due to few number of patient at this time point

6. Secondary Outcome: Time to Definitive Deterioration of the FKSI-DRS Risk Score by at Least 3 Score Units by First-line Drug
Description: The Functional Assessment of Cancer Therapy - Kidney Symptom Index, Disease Related Symptoms (FKSI-DRS) is a set of items to assess symptoms experienced by patients with advanced kidney cancer. These symptoms include fatigue, pain, weight loss, dyspnea, cough, fever and hematuria. Each item is scored on a 5-point scale (0 = not at all; 4 = very much). The FKSI-DRS total score ranges from 0 (most severe symptoms) to 36 (no symptoms). Definitive deterioration was defined as a decrease by at least 3 units compared to baseline, with no later increase above this threshold observed during the 1-L of treatment. A single measure reporting a decrease of at least 3 units was considered definitive only if it was the last one available for the patient.
Time Frame: <=14 days prior to the first dose of study medication, on day 1, day 28 of every cycle, at the end of treatment visit, at the 28 day FUP visit and monthly thereafter for up to 3 months or until initiation of another anticancer therapy up to 35 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus 1L/Sunitinib 2L | Sunitinib 1L/Everolimus 2L
Number analyzed (Participants) | 238 | 233
Months | 12.65 [7.9 to 19.4] | 16.66 [13.7 to NA] — N/A = Data not estimable due to few number of patient at this time point

7. Secondary Outcome: Time to Definitive Deterioration of the FKSI-DRS Risk Score by at Least 3 Score Units by First and Second-line Drugs Combined
Description: The Functional Assessment of Cancer Therapy - Kidney Symptom Index, Disease Related Symptoms (FKSI-DRS) is a set of items to assess symptoms experienced by patients with advanced kidney cancer. These symptoms include fatigue, pain, weight loss, dyspnea, cough, fever and hematuria. Each item is scored on a 5-point scale (0 = not at all; 4 = very much). The FKSI-DRS total score ranges from 0 (most severe symptoms) to 36 (no symptoms). Definitive deterioration was defined as a decrease by at least 3 units compared to baseline, with no later increase above this threshold observed during the 1-L or 2-L treatment. A single measure reporting a decrease of at least 3 units was considered definitive only if it was the last one available for the patient.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus 1L/Sunitinib 2L | Sunitinib 1L/Everolimus 2L
Number analyzed (Participants) | 238 | 233
Months | 14.23 [12.0 to 19.4] | 15.97 [13.7 to 20.4]

8. Secondary Outcome: Time to Definitive Deterioration of the Physical Functioning (PF) Scale of the EORTC QLQ-C30 - by First-Line (1L) Drug
Description: The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) contains 30 items. These include a global health status/QoL scale, five functional scales, three symptom scales, and six single items. The standardized score for the PF, fatigue subscales and global health status ranges from 0 to 100, with a higher score representing a high level of functioning/high level of symptom/high quality of life. Definitive deterioration by at least 10% was defined as a decrease in score by at least 10% compared to baseline, with no later increase above this threshold observed during the first line of treatment. A single measure reporting a decrease of at least 10% was considered definitive only if it was the last one available for the participant.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus 1L/Sunitinib 2L | Sunitinib 1L/Everolimus 2L
Number analyzed (Participants) | 238 | 233
Months | 13.47 [7.9 to 20.6] | 14.03 [12.1 to 17.7]

9. Secondary Outcome: Time to Definitive Deterioration of the Physical Functioning Scale of the EORTC QLQ-C30 - by First and Second-Line Drugs Combined
Description: The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) contains 30 items. These include a global health status/QoL scale, five functional scales, three symptom scales, and six single items.The standardized score for the PF, fatigue subscales and global health status ranges from 0 to 100, with a higher score representing a high level of functioning/high level of symptom/high quality of life. Definitive deterioration by at least 10% was defined as a decrease in score by at least 10% compared to baseline, with no later increase above this threshold observed during the first line or second line treatment. A single measure reporting a decrease of at least 10% was considered definitive only if it was the last one available for the participant.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus 1L/Sunitinib 2L | Sunitinib 1L/Everolimus 2L
Number analyzed (Participants) | 238 | 233
Months | 12.25 [9.5 to 16.3] | 14.03 [12.0 to 17.7]

10. Secondary Outcome: Time to Definitive Deterioration of the Global Health Status/QoL Scores of the EORTC QLQ-C30 by First-Line Drug
Description: The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) contains 30 items. These include a global health status/QoL scale, five functional scales, three symptom scales, and six single items.The standardized score for the PF, fatigue subscales and global health status ranges from 0 to 100, with a higher score representing a high level of functioning/high level of symptom/high quality of life. Definitive deterioration by at least 10% was defined as a decrease in score by at least 10% compared to baseline, with no later increase above this threshold observed during the first line of treatment. A single measure reporting a decrease of at least 10% was considered definitive only if it was the last one available for the participant.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus 1L/Sunitinib 2L | Sunitinib 1L/Everolimus 2L
Number analyzed (Participants) | 238 | 233
Months | 7.92 [5.6 to 12.1] | 12.25 [7.9 to 14.1]

11. Secondary Outcome: Time to Definitive Deterioration of the Global Health Status/QoL Scores of the EORTC QLQ-C30 by First and Second-Line Drugs Combined
Description: The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) contains 30 items. These include a global health status/QoL scale, five functional scales, three symptom scales, and six single items. The standardized score for the PF, fatigue subscales and global health status ranges from 0 to 100, with a higher score representing a high level of functioning/high level of symptom/high quality of life. Definitive deterioration by at least 10% was defined as a decrease in score by at least 10% compared to baseline, with no later increase above this threshold observed during the first line or second line treatment. A single measure reporting a decrease of at least 10% was considered definitive only if it was the last one available for the participant.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus 1L/Sunitinib 2L | Sunitinib 1L/Everolimus 2L
Number analyzed (Participants) | 238 | 233
Months | 10.84 [7.5 to 13.8] | 12.71 [10.5 to 14.8]

12. Secondary Outcome: Time to Definitive Deterioration of the Fatigue Scale of the EORTC QLQ-C30 by First-Line Drug
Description: as for outcome 10
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus 1L/Sunitinib 2L | Sunitinib 1L/Everolimus 2L
Number analyzed (Participants) | 238 | 233
Months | 9.20 [6.2 to 12.6] | 11.37 [9.3 to 13.4]

13. Secondary Outcome: Time to Definitive Deterioration of the Fatigue Scale of the EORTC QLQ-C30 by First and Second-Line Drugs Combined
Description: as for outcome 11
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Everolimus 1L/Sunitinib 2L | Sunitinib 1L/Everolimus 2L
Number analyzed (Participants) | 238 | 233
Months | 11.56 [7.9 to 14.1] | 13.34 [10.8 to 15.9]

ADVERSE EVENTS:
Arm/Group | Everolimus 1L/Sunitinib 2L | Sunitinib 1L/Everolimus 2L
Serious Adverse Events (participants affected / at risk) | 139/238 | 131/231
Other Adverse Events (participants affected / at risk) | 231/238 | 228/231
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus 1L/Sunitinib 2L (N=238) | Sunitinib 1L/Everolimus 2L (N=231)
Anaemia (Blood and lymphatic system disorders) | 16 | 9
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 9
Acute myocardial infarction (Cardiac disorders) | 1 | 2
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 7 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 3 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 2
Myocardial infarction (Cardiac disorders) | 3 | 3
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 2 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular dysfunction (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 2
Corneal disorder (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 8
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1
Anal fissure (Gastrointestinal disorders) | 2 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 2 | 2
Colitis (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 6 | 5
Diverticulum (Gastrointestinal disorders) | 1 | 0
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal erosion (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 2
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 3 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 3 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 4 | 5
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 3 | 0
Peritoneal adhesions (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 6 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 8
Asthenia (General disorders) | 6 | 6
Fatigue (General disorders) | 6 | 5
General physical health deterioration (General disorders) | 3 | 4
Generalised oedema (General disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 1
Influenza like illness (General disorders) | 1 | 1
Localised oedema (General disorders) | 0 | 1
Malaise (General disorders) | 3 | 1
Mucous membrane disorder (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 2 | 3
Oedema peripheral (General disorders) | 2 | 3
Pelvic mass (General disorders) | 0 | 1
Performance status decreased (General disorders) | 1 | 1
Peripheral swelling (General disorders) | 1 | 2
Pyrexia (General disorders) | 10 | 7
Sudden death (General disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 4
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Haemobilia (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1
Abscess oral (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Aspergillus infection (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bacterial prostatitis (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 3 | 3
Clostridium difficile infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 2
Empyema (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 1
Hepatitis A (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infected bites (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 18 | 15
Respiratory tract infection (Infections and infestations) | 2 | 0
Salmonella sepsis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 4
Septic shock (Infections and infestations) | 4 | 2
Urinary tract infection (Infections and infestations) | 3 | 5
Wound infection (Infections and infestations) | 1 | 0
Wound sepsis (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 2
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 3 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Scar (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 3 | 3
Body temperature increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 1
Eastern cooperative oncology group performance status worsened (Investigations) | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 2
Hepatic enzyme increased (Investigations) | 0 | 1
Troponin (Investigations) | 0 | 1
Troponin I increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 13 | 6
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1
Feeding disorder (Metabolism and nutrition disorders) | 1 | 0
Food intolerance (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 4 | 3
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Vertebral lesion (Musculoskeletal and connective tissue disorders) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 3 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Coma (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 0
Hemiparesis (Nervous system disorders) | 2 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 2
Meningorrhagia (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 2
Somnolence (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 4 | 3
Status epilepticus (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Visual field defect (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 2
Disorientation (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 11 | 10
Anuria (Renal and urinary disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 2 | 3
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 4 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 5 | 3
Renal vein thrombosis (Renal and urinary disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 13
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Generalised erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 4
Hypertensive crisis (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 3 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus 1L/Sunitinib 2L (N=238) | Sunitinib 1L/Everolimus 2L (N=231)
Anaemia (Blood and lymphatic system disorders) | 75 | 70
Leukopenia (Blood and lymphatic system disorders) | 11 | 14
Neutropenia (Blood and lymphatic system disorders) | 21 | 45
Thrombocytopenia (Blood and lymphatic system disorders) | 37 | 58
Hyperthyroidism (Endocrine disorders) | 4 | 14
Hypothyroidism (Endocrine disorders) | 30 | 57
Periorbital oedema (Eye disorders) | 9 | 12
Abdominal discomfort (Gastrointestinal disorders) | 13 | 8
Abdominal distension (Gastrointestinal disorders) | 19 | 16
Abdominal pain (Gastrointestinal disorders) | 49 | 41
Abdominal pain upper (Gastrointestinal disorders) | 32 | 38
Aphthous stomatitis (Gastrointestinal disorders) | 14 | 2
Constipation (Gastrointestinal disorders) | 66 | 68
Diarrhoea (Gastrointestinal disorders) | 131 | 140
Dry mouth (Gastrointestinal disorders) | 16 | 22
Dyspepsia (Gastrointestinal disorders) | 37 | 59
Dysphagia (Gastrointestinal disorders) | 16 | 12
Gastritis (Gastrointestinal disorders) | 8 | 13
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 14 | 28
Mouth ulceration (Gastrointestinal disorders) | 18 | 14
Nausea (Gastrointestinal disorders) | 114 | 125
Oral pain (Gastrointestinal disorders) | 12 | 12
Stomatitis (Gastrointestinal disorders) | 134 | 146
Toothache (Gastrointestinal disorders) | 15 | 8
Vomiting (Gastrointestinal disorders) | 73 | 76
Asthenia (General disorders) | 44 | 63
Chills (General disorders) | 29 | 20
Face oedema (General disorders) | 16 | 19
Fatigue (General disorders) | 124 | 131
Non-cardiac chest pain (General disorders) | 33 | 30
Oedema peripheral (General disorders) | 79 | 58
Pain (General disorders) | 14 | 11
Peripheral swelling (General disorders) | 15 | 10
Pyrexia (General disorders) | 66 | 48
Bronchitis (Infections and infestations) | 12 | 6
Influenza (Infections and infestations) | 16 | 8
Nasopharyngitis (Infections and infestations) | 26 | 18
Pneumonia (Infections and infestations) | 16 | 10
Upper respiratory tract infection (Infections and infestations) | 25 | 38
Urinary tract infection (Infections and infestations) | 21 | 23
Alanine aminotransferase increased (Investigations) | 16 | 18
Aspartate aminotransferase increased (Investigations) | 14 | 12
Blood alkaline phosphatase increased (Investigations) | 4 | 12
Blood creatinine increased (Investigations) | 34 | 39
Gamma-glutamyltransferase increased (Investigations) | 12 | 16
Haemoglobin decreased (Investigations) | 21 | 26
Neutrophil count decreased (Investigations) | 7 | 15
Platelet count decreased (Investigations) | 6 | 17
Weight decreased (Investigations) | 63 | 49
Decreased appetite (Metabolism and nutrition disorders) | 93 | 101
Dehydration (Metabolism and nutrition disorders) | 19 | 23
Hypercholesterolaemia (Metabolism and nutrition disorders) | 19 | 12
Hyperglycaemia (Metabolism and nutrition disorders) | 41 | 30
Hyperkalaemia (Metabolism and nutrition disorders) | 12 | 14
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 21 | 15
Hypoalbuminaemia (Metabolism and nutrition disorders) | 13 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 14 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 50 | 46
Back pain (Musculoskeletal and connective tissue disorders) | 60 | 66
Bone pain (Musculoskeletal and connective tissue disorders) | 8 | 15
Flank pain (Musculoskeletal and connective tissue disorders) | 23 | 17
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 | 11
Muscular weakness (Musculoskeletal and connective tissue disorders) | 15 | 13
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 15 | 11
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 29 | 20
Myalgia (Musculoskeletal and connective tissue disorders) | 19 | 22
Neck pain (Musculoskeletal and connective tissue disorders) | 10 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 47 | 44
Dizziness (Nervous system disorders) | 40 | 30
Dysgeusia (Nervous system disorders) | 73 | 75
Headache (Nervous system disorders) | 58 | 50
Hypoaesthesia (Nervous system disorders) | 16 | 10
Neuropathy peripheral (Nervous system disorders) | 12 | 14
Paraesthesia (Nervous system disorders) | 12 | 12
Anxiety (Psychiatric disorders) | 21 | 19
Depression (Psychiatric disorders) | 22 | 13
Insomnia (Psychiatric disorders) | 41 | 41
Dysuria (Renal and urinary disorders) | 19 | 15
Haematuria (Renal and urinary disorders) | 12 | 17
Proteinuria (Renal and urinary disorders) | 6 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 96 | 76
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 13 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 68 | 57
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 18 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 53 | 54
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 28 | 22
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 14 | 11
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 16 | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 24 | 19
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 26 | 17
Alopecia (Skin and subcutaneous tissue disorders) | 15 | 15
Dermatitis (Skin and subcutaneous tissue disorders) | 4 | 12
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 20 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 34 | 38
Erythema (Skin and subcutaneous tissue disorders) | 11 | 18
Hair colour changes (Skin and subcutaneous tissue disorders) | 6 | 16
Nail disorder (Skin and subcutaneous tissue disorders) | 13 | 10
Night sweats (Skin and subcutaneous tissue disorders) | 9 | 13
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 46 | 92
Pruritus (Skin and subcutaneous tissue disorders) | 43 | 38
Rash (Skin and subcutaneous tissue disorders) | 95 | 67
Swelling face (Skin and subcutaneous tissue disorders) | 12 | 6
Yellow skin (Skin and subcutaneous tissue disorders) | 12 | 28
Hypertension (Vascular disorders) | 61 | 84

LIMITATIONS AND CAVEATS:
PRO Tools - completed on Days 1 & 28 of a cycle. Assessments on D1 coincided with end of a 14-day break for patients on sunitinib but not everolimus. So D1 assessments of patients in sunitinib arm may be less impacted by potential toxicity effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.